CLINICAL TRIAL: NCT01685879
Title: Glycemic Response to High Amylose Rice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Principal Investigator, Maria Stewart, Assistant Professor, University of Hawaii
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HARice; Project HAW00262H (Other Grant/Funding Number: USDA)
Record Dates: First submitted 2012-09-11; First posted 2012-09-14 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Treatment (Pilot Study)
Keywords: postprandial glycemic response; postprandial insulin response; rice; appetite; hunger

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- High Amylose Rice 1 (Experimental): Test rice with high dietary fiber content
  Interventions: Other: Rice
- High Amylose Rice 2 (Experimental): Test rice with high dietary fiber content
  Interventions: Other: Rice
- Control Rice (Placebo Comparator): Rice portion that contains 50 g carbohydrate.
  Interventions: Other: Rice
- Glucose beverage (Placebo Comparator): Glucose beverage with 50 g carbohydrate
  Interventions: Other: Glucose Beverage

INTERVENTIONS:
Other: Rice — Rice portion containing 50 g total carbohydrate
  Arms: High Amylose Rice 1
Other: Rice — Rice portion that provides 50 g total carbohydrate.
  Arms: High Amylose Rice 2
Other: Rice — Rice portion that provides 50 g total carbohydrate.
  Arms: Control Rice
Other: Glucose Beverage — Glucose beverage that provides 50 g total carbohydrate.
  Arms: Glucose beverage

SUMMARY:
Certain types of rice have more dietary fiber than others. This type of rice is known a "high amylose rice." This study hypothesizes that high-amylose rice, will decrease blood glucose and insulin responses after consumption compared to conventional rice in healthy adults, ages 18-40. Eighteen healthy men and women will participate in this study. This study will determine how high blood glucose and insulin values rise after eating a portion of rice. This study will also evaluate hunger ratings after consuming rice. The results of this study will help researchers better understand how diet can influence diabetes management.

DETAILED DESCRIPTION:
This is a pilot study to assess glucose response in humans to a rice sample prepared with high amylose rice (high amylose rice 1 and high amylose rice 2), compared to conventional rice and a glucose test beverage.

Study Design: The proposed study is a randomized single-blind crossover design with repeated measures using human subjects (clinical study).

Treatment: The amount of resistant starch, a type of dietary fiber, is greater for high amylose varieties of rice than conventional varieties of rice. High amylose rice is commercially produced in Louisiana and Arkansas, USA. This specific rice has been bred to contain more amylose than ordinary (conventional) rice. This food is not genetically modified.

Brief Methods: Study subjects (men and women) aged 18-40 years old will be recruited from the UH-Manoa campus and Honolulu area via flyers. Interested individuals will be screened by telephone for initial eligibility (nonsmoker, non-vegetarian, habitual breakfast eater, able to fast for 12 hours, available 7:00am-10:00 am on weekdays, willing to participate in study). Based on the initial phone screening, eligible study subjects will attend an enrollment visit to complete the consent form, obtain study materials, and confirm health status and eligibility based on subject inclusion and exclusion criteria. Individuals who do not meet study eligibility will have all records destroyed. 18 healthy subjects (9 men and 9 women) will attend 4 morning study visits at the RMATRIX CRC at The Queens Medical Center. Subjects will complete a 24-hour food record for the 24 hours prior to the study visit. Subjects will be fasted for 12 hours at the time of the study visit. Upon arrival, subjects will have an IV inserted for serial blood draws, fasting blood samples will be obtained (time = 0). Subjects will then be presented one of four treatments in random order: high amylose rice-1, high amylose rice-2, conventional rice or glucose beverage. Subjects will be instructed to consume the sample or beverage within 15 minutes. Blood samples will be taken at 15, 30, 45, 60, 90, and 120 minutes. Subjects will complete an appetite survey after each blood draw. Upon completion of the study visit, subjects will be offered a snack and juice and monitored for safety.

Study staff: A graduate research assistant in the Nutrition graduate program will coordinate the clinical study. Undergraduate research assistants will assist with study visits. All students will be working under Dr. Stewart's supervision. All study staff will complete UHM biosafety training, UMH blood borne pathogens training, and UMH or NIH human subjects training.

Clinical Support: The study will be supported by nursing staff from the RMATRIX PCR to perform IV catheter insertion, collect serial blood samples and monitor for adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male or female

  * Age 18-40 years old
  * In good general health
  * Habitual breakfast eater
  * Able to fast for 12 hours
  * Available 7:00am-9:30am on weekdays
  * Willing to participate in study and complete 4 study visits within a 6-week period
  * Capable of giving informed consent

Exclusion Criteria:

* Current smoker
* BMI > 30 kg/m2
* Current use of medications that alter appetite (antidepressants, antibiotics, weight loss medications, or appetite suppressants)
* Current use of medications to control blood glucose, insulin or insulin receptors
* History of pre-diabetes, diabetes, hyperglycemia, hyperinsulinemia, gastrointestinal disease or surgery, or eating disorders
* Food allergy of any kind
* Vegetarian
* For females, pregnancy (current or within past 6 months) or lack of a regular menstrual cycle.
* History of bleeding or clotting disorders (e.g. hemophilia, thrombocytopenia, Vitamin K deficiency, liver failure)
* Current use of medications or supplements that may interfere with clotting and prolong bleeding time (e.g. aspirin, NSAIDS, coumadin, other anticoagulant therapy, herbal supplements including, but not limited to curcumin and flavonoids)
* Problems with vascular access or difficulty tolerating blood draws

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Blood Glucose response | 120 minutes
  Evaluated changes in blood glucose after consuming a bolus of carbohydrate from rice or a standard glucose beverage.

SECONDARY OUTCOMES:
Insulin Response | 120 minutes
  Measure insulin concentrations after consuming a bolus of carbohydrate from rice or standard glucose beverage.
Appetite Response | 120 minutes
  Measure appetite after consuming a bolus of carbohydrate from rice or standard glucose beverage.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Stewart, PhD, Principal Investigator — University of Hawaii at Manoa
Locations (1):
- University of Hawaii at Manoa, Honolulu, Hawaii, United States